CLINICAL TRIAL: NCT00581217
Title: A Randomized Comparison Study of Aquacel Ag and Glucan II as Donor Site Dressings With Regards to Healing Time, Cosmesis, Infection Rate, and Patient's Perceived Pain: a Pilot Study.
Brief Title: A Randomized Comparison Study of Aquacel Ag and Glucan II as Donor Site Dressings
Status: Terminated | Type: Observational
Why Stopped: Study Investigator has suddenly died, study has no results.
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-4881
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Burns
Keywords: Burn injury; Skin graft; Donor site dressing; Outcomes; Infection rate; Healing time; Cosmetic Result; Pain; Burn injured patients requiring skin grafting
MeSH Terms: conditions — Burns; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single arm study: Burn patients or patients with skin loss requiring split-thickness skin graft
  Interventions: Other: Aquacel Ag; Other: Glucan II

INTERVENTIONS:
Other: Aquacel Ag — Aquacel Ag will be applied to one donor site.
Other: Glucan II — Glucan II to be applied to a donor site on same patient for comparison

SUMMARY:
The research will be looking at patient outcomes for healing of donor sites after a split-thickness skin graft procedure for a burn or skin tissue loss. Donor site healing time, infection rate, cosmetic outcome, and patient's rating of pain will be compared between two donor site dressings, Glucan II and Aquacel Ag.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age 18 who have sustained a 1 - 30% total body surface area burn or skin tissue loss and require skin grafting

Exclusion Criteria:

* Individuals under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Burn injured patients or patients who have had full thickness skin loss requiring skin grafting and donor site dressings
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-12; Primary Completion 2010-03 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Healing time | 7 - 14 days

SECONDARY OUTCOMES:
Infection rate | 1-21 days
Cosmetic outcome | 6 months
Pain rating | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marianne E Cinat, MD, Principal Investigator — University of California, Irvine; Suzanne Bailey, PT, Principal Investigator — University of California, Irvine; Melissa Carmean, PT, CWS, BS, Principal Investigator — University of California, Irvine
Locations (1):
- University of California Irvine Medical Center, Orange, California, United States